CLINICAL TRIAL: NCT07157696
Title: Advanced Bedside Lung Imaging and Respiratory Muscle Monitoring for Respiratory Support Management in Chronically Ill Patients With Acute Respiratory Failure: From Hospital to Home
Brief Title: Advanced Respiratory Monitoring and Oxygen Therapy in Chronically Ill Patients With Acute Respiratory Failure
Acronym: HOME- Oxygen
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: Arcispedale S. Anna, Ferrara (Unknown); University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Professor, Università degli Studi di Ferrara
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HOME- Oxygen Trial
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Chronic Respiratory Failure; Cardiac Disease, Pulmonary Disease; Acute Respiratory Failure (ARF)
MeSH Terms: conditions — Heart Diseases; Lung Diseases | interventions — Oxygen Inhalation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow nasal cannulae treatment (Experimental): Participants assigned to this arm will receive home-based high-flow nasal cannula (HFNC) oxygen therapy using the myAirvo™3 device. The device delivers warm, humidified air with supplemental oxygen at a flow rate of ≥30 liters per minute, set at 37°C. Oxygen will be adjusted to maintain blood oxygen saturation (SpO₂) at or above 92%.
  • Group HFNC will receive HFNC during weeks 1-2, followed by a 2-day washout period, then low-flow oxygen during weeks 3-4, followed by a second 2-day washout period, and will resume HFNC during weeks 5-6
  Interventions: Device: High-Flow Nasal Cannula (HFNC) Oxygen Therapy; Device: Oxygen therapy
- Oxygen low therapy (Active Comparator): Participants assigned to this arm will receive standard long-term oxygen therapy delivered by a conventional low-flow oxygen device. Oxygen will be titrated to maintain blood oxygen saturation (SpO₂) at or above 92%. • Group low flow oxygen will receive low-flow oxygen during weeks 1-2, followed by a 2-day washout period, then HFNC during weeks 3-4, followed by a second 2-day washout period, and will resume low-flow oxygen during weeks 5-6.
  Interventions: Device: High-Flow Nasal Cannula (HFNC) Oxygen Therapy; Device: Oxygen therapy

INTERVENTIONS:
Device: High-Flow Nasal Cannula (HFNC) Oxygen Therapy — Type: Device / Procedure
  Description: Humidified high-flow nasal cannula oxygen therapy delivered via a home device. Provides warmed (37°C), humidified air and supplemental oxygen at ≥30 L/min, titrated to maintain oxygen saturation (SpO₂) ≥92%. Patients are instructed to use the device for ≥8 hours per day, preferably overnight.
  Special Features: Integrated remote monitoring system that automatically records flow, FiO₂, SpO₂, heart rate, and usage time, transmitting data to a secure cloud platform for clinical follow-up.
Device: Oxygen therapy — Type: Device / Procedure
  Description: Standard long-term oxygen therapy delivered through conventional low-flow systems (e.g., nasal cannula or mask). Oxygen is titrated to maintain oxygen saturation (SpO₂) ≥92%. Patients are instructed to use oxygen for ≥8 hours per day, preferably overnight.
  Special Features: No humidification, high-flow delivery, or remote monitoring capabilities.

SUMMARY:
This study is testing whether a new type of home oxygen therapy, called high-flow nasal cannula (HFNC), can improve breathing comfort and quality of life for people with long-term lung or heart conditions who need oxygen after leaving the hospital.

HFNC delivers warm, humidified oxygen at higher flow rates than standard oxygen therapy, which may reduce shortness of breath, improve sleep, and make daily activities easier. The therapy will be provided using the myAirvo™3 device, which also allows doctors to check patients' oxygen levels, heart rate, and symptoms remotely. All patients will also wear a small device (RootiREX) to monitor heart rhythm, sleep quality, and detect breathing pauses at night.

Participants will try both treatments - HFNC and standard oxygen therapy - for short periods, in random order, so that researchers can directly compare the effects within the same patient. Each treatment period will last two weeks, with a short break in between.

The main goal of the study is to see whether HFNC reduces shortness of breath (measured by the modified Medical Research Council scale). Other outcomes include comfort, sleep quality, quality of life, oxygen levels, and how well patients are able to use the devices at home.

The study will last six weeks in total for each participant. Researchers expect that HFNC will improve breathing comfort, stabilize oxygen levels, and reduce the need for hospital visits during this time.

ELIGIBILITY:
Inclusion Criteria: Adults (≥18 years) with chronic respiratory (e.g., COPD, interstitial lung disease) and/or cardiac disease (e.g., heart failure), Clinical indication for long-term oxygen therapy, Capability to manage home-based devices independently or with caregiver assistance Signed informed consent

Exclusion Criteria:

Life expectancy < 3 months Inability to comply with home follow-up procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-10-03 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
dyspnea modification | Change from the enrollment in the study to 6 weeks
  Change from the enrollment in the study to 6 weeks in dyspnea level measured by the modified Medical Research Council (mMRC) scale

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nagata K, Kikuchi T, Horie T, Shiraki A, Kitajima T, Kadowaki T, Tokioka F, Chohnabayashi N, Watanabe A, Sato S, Tomii K. Domiciliary High-Flow Nasal Cannula Oxygen Therapy for Patients with Stable Hypercapnic Chronic Obstructive Pulmonary Disease. A Multicenter Randomized Crossover Trial. Ann Am Thorac Soc. 2018 Apr;15(4):432-439. doi: 10.1513/AnnalsATS.201706-425OC. PMID 29283682
- [Result] Weinreich UM, Burchardt C, Huremovic J. The effect of domiciliary high flow nasal cannula treatment on dyspnea and walking distance in patients with interstitial lung disease - A pilot study. Chron Respir Dis. 2022 Jan-Dec;19:14799731221137085. doi: 10.1177/14799731221137085. PMID 36366859